CLINICAL TRIAL: NCT00960141
Title: A Multicenter, Double-Blind, Randomized, Parallel-Group Study Investigating the Clinical Effect of Montelukast in Patients With Seasonal Allergic Rhinitis-Fall Study
Brief Title: A Study Investigating the Effect of Montelukast in Patients With Seasonal Allergic Rhinitis (MK-0476-192)(COMPLETED)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0476-192; MK0476-192; 2009_633
Record Dates: First submitted 2009-08-14; First posted 2009-08-17 (Estimated); Results first posted 2010-06-09 (Estimated); Last update posted 2022-02-03 (Actual); Status verified 2022-02

CONDITIONS: Seasonal Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal | interventions — montelukast

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): montelukast
  Interventions: Drug: montelukast sodium
- 2 (Active Comparator): loratadine
  Interventions: Drug: Comparator: loratadine
- 3 (Placebo Comparator): placebo
  Interventions: Drug: Comparator: placebo

INTERVENTIONS:
Drug: montelukast sodium — montelukast 10 mg tablet, taken orally once daily at bed time for 2 weeks
  Arms: 1
Drug: Comparator: loratadine — loratadine 10 mg tablet, taken orally once daily at bed time for 2 weeks
  Arms: 2
Drug: Comparator: placebo — placebo tablet, taken orally once daily at bed time for 2 weeks
  Arms: 3

SUMMARY:
A study of the ability of montelukast to improve signs and symptoms of seasonal allergic rhinitis compared with placebo. Loratadine is included in the study as an active control.

ELIGIBILITY:
Inclusion Criteria:

* Patient has a documented clinical history of seasonal allergic rhinitis symptoms that become worse during the study season
* Patient is a non-smoker
* Patient is in good mental and physical health

Exclusion Criteria:

* Patient is hospitalized
* Patient is a woman who is <8 weeks postpartum or is breast feeding
* Patient intends to move or vacation away during the study
* Patient is a current or past abuser of alcohol or illicit drugs

Ages: 15 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 829 (Actual)
Dates: Start 2000-08; Primary Completion 2000-10 (Actual); Study Completion 2000-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Result] Chervinsky P, Philip G, Malice MP, Bardelas J, Nayak A, Marchal JL, van Adelsberg J, Bousquet J, Tozzi CA, Reiss TF. Montelukast for treating fall allergic rhinitis: effect of pollen exposure in 3 studies. Ann Allergy Asthma Immunol. 2004 Mar;92(3):367-73. doi: 10.1016/S1081-1206(10)61576-1. PMID 15049402

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Twenty-nine study centers in the United States.
  Therapy Period: August 2000 to October 2000
Pre-assignment Details: Patients who required excluded medication and those who did not meet a minimum predefined level of combined daytime nasal symptoms score during the run-in period were excluded from randomization.
Groups:
- Placebo: Montelukast matching-image and Loratadine matching-image placebo tablets orally once daily at bedtime for 2 weeks
- Montelukast: Montelukast 10 mg tablet and Loratadine matching-image placebo tablet orally once daily at bedtime for 2 weeks.
- Loratadine: Montelukast matching-image placebo tablet and Loratadine 10 mg tablet orally once daily at bedtime for 2 weeks.
Period: Overall Study
Arm/Group | Placebo | Montelukast | Loratadine
Started | 333 | 326 | 170
Completed | 323 | 309 | 163
Not Completed | 10 | 17 | 7
Not completed — Adverse Event | 4 | 8 | 2
Not completed — Lack of Efficacy | 3 | 4 | 2
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Protocol Violation | 1 | 3 | 2
Not completed — Withdrawal by Subject | 1 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Montelukast | Loratadine | Total
Number analyzed (Participants) | 333 | 326 | 170 | 829
Age, Continuous [Mean (Full Range); unit: years] | 36.4 [15 to 82] | 36.3 [15 to 75] | 37.5 [15 to 66] | 36.6 [15 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 222 | 227 | 119 | 568
  Male | 111 | 99 | 51 | 261
Daytime Eye Symptoms score [Mean (Standard Deviation); unit: Units on a Scale] — Patients were asked to rate each eye symptom (tearing, itchy, red, and puffy eyes) daily in the evening on a 4-point scale [0(best) to 3(worst)]. The Daytime Eye Symptoms score is the average of these 4 symptoms. Baseline is computed as average of daily values during the prerandomization run-in period.
  Units on a Scale | 1.46 (0.78) | 1.46 (0.76) | 1.44 (0.80) | 1.46 (0.77)
Daytime Nasal Symptoms Score [Mean (Standard Deviation); unit: Units on a Scale] — Patients were asked to rate each of 4 nasal symptoms (Congestion, Rhinorrhea, Itching, and Sneezing) daily in the evening on a 4-point scale [0(best) to 3(worst)]. The Daytime Nasal Symptoms Score is the average of these 4 symptoms . Baseline is computed as average of daily values during the prerandomization run-in period (includes the 3 to 5 days prior to Visit 3).
  Units on a Scale | 2.09 (0.44) | 2.14 (0.43) | 2.08 (0.40) | 2.11 (0.43)
Nighttime Symptoms Score [Mean (Standard Deviation); unit: Units on a Scale] — Patients were asked to rate each symptom (Nasal Congestion Upon Awakening, Difficulty Going to Sleep, and Nighttime Awakenings) daily in the morning on a 4-point scale [0(best) to 3(worst)]. The Nighttime Symptoms Score is the average of these 3 symptoms. Baseline is computed as average of daily values during the prerandomization run-in period.
  Units on a Scale | 1.53 (0.62) | 1.49 (0.60) | 1.54 (0.68) | 1.52 (0.62)
Rhinoconjunctivitis Quality-of-Life score [Mean (Standard Deviation); unit: Units on a Scale] — Patients completed a validated, self-administered Rhinoconjunctivitis Quality-of-Life Questionnaire Scored [0(best) to 3(worst)].
  Units on a Scale | 3.18 (1.00) | 3.20 (1.00) | 3.26 (1.08) | 3.20 (1.02)

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Daytime Nasal Symptoms Score
Description: Mean change from baseline in Daytime Nasal Symptoms score on a 4-point scale [0(best) to 3(worst)]. The average of the 4 individual nasal symptoms scores (Congestion, Rhinorrhea, Itching, and Sneezing) was reported as the Daytime Nasal Symptoms Score.
Time Frame: Baseline and Week 2
Population: The primary efficacy analyses were based on the intention-to-treat (all-patients-treated) principle, i.e., all patients who had a baseline and at least one posttreatment measurement were included.
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a Scale
Arm/Group | Placebo | Montelukast | Loratadine
Number analyzed (Participants) | 331 | 326 | 163
Units on a Scale | -0.32 [-0.37 to -0.26] | -0.38 [-0.44 to -0.32] | -0.47 [-0.55 to -0.39]

2. Secondary Outcome: Mean Change From Baseline in Nighttime Symptoms Score
Description: Mean change from baseline in Nighttime Symptoms Score on a 4-point scale [0(best) to 3(worst)]. The average of 3 scores (Nasal Congestion Upon Awakening, Difficulty Going to Sleep, and Nighttime Awakenings) was reported as the Nighttime Symptoms Score.
Time Frame: Baseline and Week 2
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a Scale
Arm/Group | Placebo | Montelukast | Loratadine
Number analyzed (Participants) | 331 | 326 | 163
Units on a Scale | -0.18 [-0.23 to -0.13] | -0.28 [-0.33 to -0.23] | -0.26 [-0.34 to -0.19]

3. Secondary Outcome: Mean Change From Baseline in Daytime Eye Symptoms Score
Description: Mean change from baseline in Daytime Eye Symptoms scores on a 4-point scale [0(best) to 3(worst)]. The average of the 4 individual eye symptoms scores (tearing, itchy, red, and puffy eyes) was reported as the Daytime Eye Symptoms Score.
Time Frame: Baseline and Week 2
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a Scale
Arm/Group | Placebo | Montelukast | Loratadine
Number analyzed (Participants) | 331 | 326 | 163
Units on a Scale | -0.23 [-0.28 to -0.17] | -0.29 [-0.35 to -0.24] | -0.35 [-0.43 to -0.28]

4. Secondary Outcome: Patient's Global Evaluation of Allergic Rhinitis
Description: An evaluation by the patient, administered at the last visit (or upon discontinuation) using a 7-point scale, in answer to a single question regarding the change in symptoms as compared to the beginning of the study. Responses were assigned numerical values from 0 (very much better) to 6 (very much worse).
Time Frame: Week 2 (or upon discontinuation)
Population: The primary efficacy analyses were based on the intention-to-treat. Since only 1 measurement was obtained during the treatment period, no missing values were imputed.
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a Scale
Arm/Group | Placebo | Montelukast | Loratadine
Number analyzed (Participants) | 333 | 324 | 169
Units on a Scale | 2.62 [2.45 to 2.78] | 2.43 [2.26 to 2.60] | 2.27 [2.04 to 2.50]

5. Secondary Outcome: Physician's Global Evaluation of Allergic Rhinitis
Description: An evaluation by the physician, administered at the last visit (or upon discontinuation) using a 7-point scale, of the change in symptoms as compared to the beginning of the study. Responses were assigned numerical values from 0 (very much better) to 6 (very much worse).
Time Frame: Week 2
Population: as for outcome 4
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a Scale
Arm/Group | Placebo | Montelukast | Loratadine
Number analyzed (Participants) | 331 | 324 | 169
Units on a Scale | 2.53 [2.38 to 2.68] | 2.35 [2.20 to 2.50] | 2.26 [2.05 to 2.46]

6. Secondary Outcome: Mean Change From Baseline in Rhinoconjunctivitis Quality-of-Life Score
Description: Patients completed a validated, self-administered questionnaire, which included 28 questions on a 7-point scale [score 0 (best) to 6 (worst)] across 7 domains: activities, sleep, non-nose/eye symptoms, practical problems, nasal symptoms, eye symptoms, and emotional. The scores for each domain were averaged, then the scores for the 7 domains were averaged for the overall score.
Time Frame: Baseline and Week 2
Population: The primary efficacy analyses were based on the intention-to-treat (all-patients-treated) principle, i.e., all patients who had a baseline and at least one posttreatment measurement were included. No missing values were imputed.
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a Scale
Arm/Group | Placebo | Montelukast | Loratadine
Number analyzed (Participants) | 330 | 324 | 168
Units on a Scale | -0.75 [-0.86 to -0.63] | -0.85 [-0.96 to -0.73] | -0.97 [-1.13 to -0.82]

ADVERSE EVENTS:
Time Frame: Over the 2-week treatment period and including 14 days follow-up post-treatment
Arm/Group | Placebo | Montelukast | Loratadine
Serious Adverse Events (participants affected / at risk) | 0/333 | 1/326 | 0/170
Other Adverse Events (participants affected / at risk) | 19/333 | 13/326 | 8/170
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=333) | Montelukast (N=326) | Loratadine (N=170)
Depression (Psychiatric disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=333) | Montelukast (N=326) | Loratadine (N=170)
Headache (Nervous system disorders) | 19 | 13 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.